CLINICAL TRIAL: NCT04362579
Title: Advanced Multi-Modal Wearable Sensing for the Prediction of Pre-Term Labor
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: STU00210698
Record Dates: First submitted 2020-04-15; First posted 2020-04-27 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy Preterm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects seen in hospital: Subjects will be recruited from Prentice Women's Hospital inpatient antepartum and labor and delivery services, and the outpatient Obstetrics and Gynecology practice, located within Galter tower with the assistance of staff.
  Interventions: Device: wearable vital signs sensor
- Home Study subjects: Subjects will be prescreened by an IRB approved staff and recruited from Prentice Women's Hospital's Department of Obstetrics and Gynecology.
  Interventions: Device: wearable vital signs sensor

INTERVENTIONS:
Device: wearable vital signs sensor — vital signs monitoring during maternal non-stress testing or in the home setting

SUMMARY:
Percent agreement of vital signs monitoring between the experimental sensor and standard of care monitoring

DETAILED DESCRIPTION:
The primary objective of the Prentice study is to assess and validate EMG performance of the new home-use sensor with extended battery life in detecting continuous EHG in a range of uterine contraction intensities, frequencies, and durations compared to gold-standard FDA-cleared tocodynamometer (GE Corometrics 250cx) in non-stress testing for antepartum surveillance.

An "at-home" study will validate the developed modifications to the wearable sensors system that provides a continuous electrohysterography (EHG) along with other additional physiological parameters (e.g. heart rate, heart rate variability, sleep quality, physical activity, and continuous blood pressure) for longitudinal monitoring in the home setting.

ELIGIBILITY:
* Maternal age >18 years old
* Pregnant mothers >13 weeks (home study only)
* Pregnant mothers >26 weeks undergoing nonstress testing or delivering
* Singleton pregnancy (inpatient or clinic visit patients only)
* History of preterm labor or premature birth, active smoker, chronic condition (ex: HTN or DM), or an interval of less than 6 months between the prior pregnancy
* Singleton pregnancy (home study only)
* No fetal abnormality or chromosomal abnormality
* Subjects willing and able to comply with requirements of the protocol

Exclusion Criteria

* Women who refuse to signed the informed consent form
* Maternal age under 18 years old
* Multiple pregnancy
* Known major fetal malformation or chromosomal abnormality
* Medical or obstetric problem that would preclude the use of abdominal electrodes
* Inability to consent to this study due to medical illness, diminished intellectual capacity, or language barrier
* Women using pacemakers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Device comparison to standard monitoring | 2 years
  The primary outcome measure is concordance of FHR tracing assessments from Rogers sensor recordings with those obtained from the current standard of care electronic fetal monitoring systems.

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xu, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States